CLINICAL TRIAL: NCT02653963
Title: Adjunctive Triamcinolone Acetonide for Ahmed Glaucoma Valve Implantation
Brief Title: Triamcinolone for Ahmed Glaucoma Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Azadeh Doozandeh, ShaheedBMU, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShaheedBMU-9467
Record Dates: First submitted 2015-12-24; First posted 2016-01-13 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Glaucoma
Keywords: Steroid, Triamcinolone, Ahmed Glaucoma valve
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional AGV (No Intervention): A limbus-based conjunctival peritomy was created 4mm posterior to the limbus and Tenon's capsule was dissected. The AGV Plate was secured to the sclera 8 mm posterior to the limbus. The tube was trimmed to an appropriate length and inserted into the anterior chamber through a corneoscleral track. The tube was fixed to the episclera with a 10-0 nylon mattress suture. A donor sclera was fashioned to cover the exposed part of the tube and was secured to the sclera using 10-0 nylon sutures. The conjunctiva and Tenon were closed using 10-0 nylon suture.
- Triamcinolone adjuctival AGV (Experimental): Subtenon Periplate 10 mg triamcinolone acetonide around the AGV plate after fixation of AGV Plate to the sclera
  Interventions: Drug: Adjunctival Triamcinolone

INTERVENTIONS:
Drug: Adjunctival Triamcinolone — Intraoperative Periplate 10 mg Triamcinolone Injection during AGV Implantation
  Other Names: Intraoperative steroid
  Arms: Triamcinolone adjuctival AGV

SUMMARY:
This triple-blind, stratified, randomized clinical trial includes 100 eyes of 100 patients aged 18 to 85 years with refractory glaucoma. Eligible subjects undergo stratified block randomization; eyes are first stratified to one of four subgroups: group 1:patients with previous failed trabeculectomy, group 2: uveitic glaucoma, group 3: neovascular glaucoma and group 4: other indications like aphakic glaucoma or glaucoma associated with vitreoretinal procedures.

In each subgroup, eyes are randomly assigned to the study arms using random blocks: conventional Ahmed Glaucoma Valve (AGV) implantation (group A, 50 eyes), Ahmed Glaucoma Valve (AGV) with intraoperative periplate triamcinolone injection (group B, 50 eyes).

Patients will be followed for one year. They will undergo full ophthalmology examination at first day, first week, month 1, 3, 6, 9 and 12 after the surgery.

The primary outcome measure is cumulative probability of success, defined as intraocular pressure (IOP) of 6-21 mm Hg, with or without medication, and no serious complications, additional glaucoma surgery, or loss of light perception.

The outcomes will be compared between two arms in each subgroup.

The number of eyes requiring medications, time to initiation of medications, and number of medications will be compared.

DETAILED DESCRIPTION:
All procedures was performed by glaucoma specialists under general anesthesia employing the same technique in all subjects. The surgical field was prepared and draped in the usual sterile fashion. After insertion of a lid speculum and irrigation with povidine iodine 5% solution, a 7-0 silk limbal traction suture was placed to rotate the globe and achieve optimal supratemporal exposure. A limbus-based conjunctival peritomy was created 4mm posterior to the limbus and Tenon's capsule was dissected using Westcott and Stevens scissors. Hemostasis was achieved using wet field bipolar cautery. The Ahmed Glaucoma Valve (AGV) plate was secured to the sclera 8 mm posterior to the limbus with two interrupted 7-0 silk sutures. The tube was trimmed to an appropriate length with the bevel facing anteriorly and inserted into the anterior chamber through a corneoscleral track created with a 23-gauge needle. The tube was fixed to the episclera with a 10-0 nylon mattress suture. A quadrangular donor scleral patch graft (4×7 mm) was fashioned to cover the exposed part of the tube and was secured to the sclera using 10-0 nylon sutures. At this stage, in adjunctive triamcinolone group, 10 mg triamcinolone was injected in the subtenon space around the Ahmed Glaucoma Valve (AGV) plate. The conjunctiva and Tenon were closed using 10-0 nylon suture in a running fashion. At the end of the procedure, a subconjunctival injection of 4 mg betamethasone and 50 mg cephazolin were given in all eyes.

All patients were examined on the first post-operative day; the postoperative regimen included topical chloramphenicol 0.5% eye drops 4 times per day for 1 week and topical betamethasone 0.1% eye drops 6 times per day which was tapered over 6 to 8 weeks, except in cases with severe inflammation which required a longer period of treatment.

Follow up examination was repeated every week during the first month and thereafter at 6 weeks, and 3, 6, 9 and 12 months after the operation. Possible complications such as endophthalmitis, choroidal effusion or hemorr, wound leakage, hyphema, hypotony, malignant glaucoma, implant exposure, tube malposition, bleb encapsulation, and decreased best corrected visual acuity (BCVA) more than 2 lines were mentioned. IOP was measured by a calibrated Goldmann applanation tonometer (SN-9007, Haag-Streit, Koniz, Switzerland). All measurements were obtained by one masked examiner.

The main outcome measure of the study was intraocular pressure and number of anti-glaucoma medications. Complete success was defined as IOP between 6 and 21 without the use of any glaucoma medication. Partial success was defined as IOP between 6 and 21 with a maximum of 2 glaucoma drops. Overall success rate was the sum of complete and partial success rates. Failure was defined as IOP>21, IOP<21 with ≥3 medications, loss of vision, shunt extrusion and need for additional glaucoma surgery. Other outcome measures included best corrected visual acuity (BCVA), number of glaucoma medications, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were patients aged 18-85 years with refractory glaucoma scheduled for AGV implantation.

Exclusion Criteria:

* Exclusion criteria was poor compliance for follow up, previous AGV implantation, concomitant procedures such as deep vitrectomy or cataract surgery, and any major intra- or postoperative complication which could affect the outcomes of surgery.
* Patients for whom AGV was implanted in any location except superior-temporal quadrant were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
INTRAOCULAR PRESSURE | 1, 3, 6 ,9 and 12 month
  Intraocular pressure (IOP) of 6-21 mm Hg, with or without medication, and no serious complication

SECONDARY OUTCOMES:
Anti-glaucoma drug number | 1, 3, 6 ,9 and 12 month
Visual acuity | 1, 3, 6 ,9 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Doozandeh, MD, Principal Investigator — Ophthalmology research center, Shahid Beheshti University Of Medical Sciences
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided